CLINICAL TRIAL: NCT05230758
Title: Phase III Randomized Double-blind Placebo-controlled Trial of Metformin for Cognitive Recovery and White Matter Growth in Paediatric Patients With a Brain Tumour
Brief Title: Effect of Metformin on Behaviour and the Brain in Children Treated for a Brain Tumour
Acronym: Met Med Can
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Donald Mabbott (Other)
Responsible Party: Sponsor-Investigator, Donald Mabbott, Psychologist, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1000073107
Record Dates: First submitted 2022-01-12; First posted 2022-02-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Medulloblastoma, Childhood; Cognitive Impairment
Keywords: Metformin; Paediatric brain tumour; Memory; Cognitive late effects
MeSH Terms: conditions — Medulloblastoma; Cognitive Dysfunction | interventions — Metformin; Tablets

STUDY DESIGN:
Intervention Model Description: We elect to employ a parallel arm superiority trial. As there is no standard of care equivalent for the intervention being investigated (i.e. metformin for improved cognition and white matter growth), a placebo is being used to prevent any potential response bias.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: We are implementing a double-blind procedure to ensure that neither participants nor members of the research team have knowledge of the randomized treatment group to prevent bias in reporting, outcome assessment and analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): Oral metformin will be administered approximately 500mg/m2/day for 1 week and increased to 1000mg/m2/day for 15 weeks. Doses will be rounded to increments of half tablets (250mg, 500mg, 750mg and 1000mg).
  Interventions: Drug: Metformin hydrochloride (HCl) 500mg tablet
- Placebo (Placebo Comparator): Oral placebo will be administered approximately 500mg/m2/day for 1 week and increased to 1000mg/m2/day for 15 weeks. Doses will be rounded to increments of half tablets (250mg, 500mg, 750mg and 1000mg).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin hydrochloride (HCl) 500mg tablet — Metformin HCl 500mg tablets contain 500mg of active pharmaceutical ingredient (API) and are white, round, biconvex, film-coated tablets, with a score line on one face and debossed with "HMR" on the other. Each tablet contains the non-medicinal ingredients magnesium stearate and povidone. Tablet coating is comprised of hydroxypropyl methylcellulose, polyethylene glycol and titanium dioxide.
  Other Names: Glucophage
  Arms: Metformin
Drug: Placebo — Matching white round tablet containing excipients only. The placebo tablets will match the active drug as closely as possible in terms of appearance.
  Other Names: Control
  Arms: Placebo

SUMMARY:
The efficacy of treatment with metformin for promoting cognitive recovery and brain growth in children/adolescents treated for a brain tumour will be investigated in a multi-site Phase III randomized double-blind placebo-controlled parallel arm superiority trial. Specifically, in children/adolescents aged 7 years to 21 years and 11 months who have completed treatment for a brain tumour, is oral administration of metformin for 16 weeks associated with greater improvement of cognitive function and brain growth compared to placebo administered for 16 weeks?

DETAILED DESCRIPTION:
A critical barrier to improving the quality of life of children/adolescents living with cancer is that our curative therapies, which include a combination of surgery, chemotherapy and radiation, have toxic effects on healthy tissue, resulting in long-term problems. This is evident for children and adolescents who survive brain tumours requiring aggressive therapy: they experience brain injury and cognitive impairment. There are few therapies for restoring cognitive function and promoting brain growth in survivors; however new work in regenerative medicine offers a possible alternative. The drug metformin promotes brain growth in animal models by activating neural stem cells. In a pilot trial with 24 participants, we found that metformin was safe and tolerable for use in children/adolescents treated with cranial radiation for a brain tumour and may improve cognition and promote white matter growth. In this multi-site clinical trial, we will test the efficacy of treatment with metformin for brain repair and cognitive recovery in paediatric medulloblastoma and other brain tumour survivors. If we find that metformin promotes cognitive improvement and brain growth in paediatric survivors of medulloblastoma and other paediatric brain tumours treated with cranial radiation, this may offer a viable therapeutic approach that may improve quality of life of these cancer patients and provide a model for treatment of late effects in other paediatric cancers.

This study is designed to test the efficacy of metformin in a 16-week multi-centre, phase III, double-blind, randomized placebo-controlled superiority trial with two parallel conditions (metformin versus placebo). Participants will be randomly assigned to one of the two treatments where they will either complete a 16-week cycle of metformin or a 16-week cycle of placebo. Participants will be randomized using Research Electronic Data Capture (REDCap) to ensure allocation concealment. The randomization code will not be released until the participant has been recruited, consented and passed screening. Outcome assessments will be conducted at Baseline immediately following the completion of week 16 treatment (Post-Intervention, Week 17), and 24 weeks following completion of the intervention (6 Month Follow-Up, Week 41).

The primary endpoint is cognitive function in children/adolescent survivors of a brain tumour at Post-Intervention (Week 17) compared to Baseline. We hypothesize that 16 weeks of treatment with metformin will be associated with better cognitive outcomes than 16 weeks of treatment with placebo. Cognitive outcomes will be measured using tests of working memory, declarative memory, and processing speed.

The key secondary outcome will be diffusion MRI within the corpus callosum at Post-Intervention (Week 17) compared to Baseline. We hypothesize that 16 weeks of treatment with metformin will be associated with increased white matter growth in the corpus callosum compared to 16 weeks of treatment with placebo. Increased white matter growth will be measured using diffusion MRI metrics.

Exploratory outcomes have been selected to investigate broader metformin-induced changes in the brain and cognition.

1. We hypothesize that 16 weeks of treatment with metformin will promote global white matter growth in the brain more so than 16 weeks of treatment with placebo at Post-Intervention (Week 17) compared to Baseline. White matter growth will be assessed using diffusion MRI metrics of myelin and fiber structure.
2. We hypothesize that 16 weeks of treatment with metformin will result in greater increases in hippocampal volume compared to that 16 weeks of treatment with placebo at Post-Intervention (Week 17) compared to Baseline. Structural MRI measures of hippocampal volume will be explored.
3. We hypothesize that 16 weeks of treatment with metformin will result in superior performance on measures of attention and executive functioning, compared to 16 weeks of treatment with placebo at Post-Intervention (Week 17) compared to Baseline. Tests of attention and executive functioning will be used.
4. We hypothesize that all outcome measures will continue in the predicted direction at 24 weeks (6 Month Follow-Up, Week 41) compared to Baseline following completion of 16 weeks of metformin compared to 16 weeks of placebo.
5. We also hypothesize that 16 weeks of treatment with metformin will yield better outcomes in females compared to males for all measures and that these findings will persist at 24 weeks (6 Month Follow-Up, Week 41) following the intervention compared to Baseline.
6. We hypothesize that 16 weeks of treatment with metformin will result in improved ratings of global health as reported by the parent/guardian at Post-Intervention (Week 17) compared to Baseline.

Metformin is a well-studied medication with a broad clinical experience in children including polycystic ovarian syndrome, diabetes, and obesity. The youngest age of use is 2 years old. The proposed dose and the schedule of administration of metformin is based on safety and toxicity data obtained from our pilot trial and previous use in paediatric populations. One hundred and twenty (120) English speaking and twenty (20) French speaking participants - aged 7 years to 21 years and 11 months - will be recruited from up to 20 sites across Canada and Australia.

Analysis of covariance (ANCOVA) will be used to examine the effects metformin versus placebo for each outcome in English speaking participants, controlling for Baseline outcome measurements. For French speaking participants, IQ testing will be completed, but not Cognitive testing as French-Canadian translations are not available. By focusing on a disease that requires some of the most aggressive therapy used in modern protocols, and by targeting the patients most vulnerable to the harmful effects of treatment we hope to provide a model of intervention that can then be applied to other cancers and actively promote brain health and cognitive recovery.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. No less than 3 weeks after completion of:

   * Primary therapy for:

     1. medulloblastoma

        OR
     2. ependymoma

        OR
     3. craniopharyngioma

        OR
     4. germ cell tumours

        OR
   * Primary therapy for any other brain tumour treated with cranial radiation - at the discretion of the Study PI

   OR
   * Cranial radiation for relapsed ependymoma
2. Age 7 years to 21 years and 11 months at the time of enrollment
3. Either declare English (or French in accepting sites) as their native language or have had at least two years of schooling in English (or French in accepting sites) at the time of consent
4. Able to swallow tablets either whole, crushed or via a feeding tube and be willing to adhere to the study intervention regimen
5. Meet criteria for normal organ function requirements as described below:

   1. Normal renal function defined as: Estimated glomerular filtration rate (eGFR) > 75ml/min/1.73m²

      * eGFR is calculated using the Schwartz formula: eGFR (mL/min/1.73m²) = (0.41 × height in cm) / creatinine in mg/dL
   2. Normal liver function defined as:

      * Serum glutamic-oxaloacetic transaminase (SGOT) (AST) ≤2.5 x institutional upper limit of normal (ULN) for age and gender
      * Serum glutamic pyruvic transaminase (SGPT) (ALT) ≤2.5 x institutional ULN for age and gender
      * Total bilirubin <1.5x institutional ULN for age and gender (patients with documented Gilbert's Disease may be enrolled with Sponsor approval and total bilirubin ≤2.0 x institutional ULN)
6. Informed consent (and assent, where applicable) will be obtained from the participants and/or their legal guardian(s) by study team members delegated to consent for this study

Exclusion Criteria:

Participants who meet any of the following criteria will not be eligible to take part in the trial:

1. Standard score of less than 60 for full scale IQ on the Wechsler Abbreviated Scale of Intelligence, Second Edition (WASI-II) (or other Wechsler Scale of Intelligence for English speaking participants) or pro-rated IQ score on the Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V) or Wechsler Adult Intelligence Scale (WAIS-IV) for French speaking participants at Screening visit
2. Have a known hypersensitivity to metformin hydrochloride
3. Have unstable and/or insulin-dependent (Type 1) diabetes
4. Have a history of hypoglycemia after 2 years of age
5. Have been diagnosed with acute or chronic metabolic acidosis and/or lactic acidosis or if bicarbonate (Total CO2) is less than 22 mmol/L at the Screening visit
6. Have a history of renal disease or renal dysfunction pre-existing to the diagnosis of Medulloblastoma
7. Have a history of congestive heart failure requiring pharmacologic treatment (including the use of diuretics) within two years prior to study entry
8. Currently taking part in a cognitive rehabilitation intervention study
9. Treatment or planned treatment involving diuretics
10. Current or planned treatment with cationic drugs excreted by the kidneys (e.g. amiloride, cimetidine, digoxin, morphine, nifedipine, procainamide, quinidine, quinine, ranitidine, triamterene, trimethoprim, and vancomycin)
11. Current or planned treatment with concomitant medications with potential unacceptable interaction with metformin including, lamotrigine, beta blockers, angiotensin-converting enzyme (ACE) inhibitors, glycopyrrolate, and carbonic anhydrase inhibitors, or at the discretion of the Site PI or delegate for medications with potential interactions such as sertraline, lansoprazole and omeprazole.
12. Pernicious anemia (according to results of the Screening visit blood draw)
13. Current use of metformin hydrochloride
14. Any condition or diagnosis, that could in the opinion of the Site PI or delegate interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study results, or put the participant at risk
15. Are receiving palliative care

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from Week 1 (Baseline) Children's Auditory Verbal Learning Test-2 (CAVLT-2)/Rey Auditory Verbal Learning Test (RAVLT) Immediate Recall at Week 17 (Post-Intervention) to Assess Declarative Memory | Week 1 (Baseline), Week 17 (Post-Intervention)
  To examine the effectiveness of 16 weeks of treatment with metformin versus 16 weeks of placebo for improving cognition, as measured by CAVLT-2/RAVLT which is a test of auditory verbal learning and memory.
Change from Week 1 (Baseline) NIH Toolbox List Sort Working Working Memory Test at Week 17 (Post-Intervention) to Assess Working Memory | Week 1 (Baseline), Week 17 (Post-Intervention)
  To examine the effectiveness of 16 weeks of treatment with metformin versus 16 weeks of placebo for improving cognition, as measured by List Sorting Working Memory Test (LSWMT) in which participants will be required to recall and place in sequence stimuli that are presented visually and verbally.
Change from Week 1 (Baseline) Cambridge Neuropsychological Test Automated Battery (CANTAB) Mean Reaction Time for Correct Trials across the RVP, RTI, MTS, and DMS Subtests at Week 17 (Post-Intervention) to Assess Processing Speed | Week 1 (Baseline), Week 17 (Post-Intervention)
  To examine the effectiveness of 16 weeks of treatment with metformin versus 16 weeks of placebo for improving cognition, as measured by mean reaction time for correct trials across subtests of the CANTAB:
  1. Rapid Visual Information Processing (RVP)
  2. Reaction Time (RTI)
  3. Match to Sample Visual Search (MTS)
  4. Delayed Matching to Sample (DMS) Each subtest provides an outcome measure of response latency, which will be averaged across all correct trials for each subtest to provide an overall measure of processing speed.

SECONDARY OUTCOMES:
Diffusion Kurtosis Imaging (DKI) to Assess White Matter Growth within the Corpus Callosum | Week 1 (Baseline), Week 17 (Post-Intervention)
  To examine the effectiveness of 16 weeks of treatment with metformin versus 16 weeks of placebo for promoting white matter growth within the corpus callosum as measured by DKI including axonal water fraction (AWF), a metric sensitive to myelin.
  This secondary outcome measure (MRI scan) was made optional to participants enrolled after April 2024.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Mabbott, Ph.D., Study Chair — The Hospital for Sick Children; Eric Bouffet, M.D., Principal Investigator — The Hospital for Sick Children
Locations (20):
- Australia (6):
  - John Hunter Children's Hospital, New Lambton Heights, New South Wales
  - Children's Hospital in Westmead, Westmead, New South Wales
  - Women and Childen's Hospital, Adelaide, North Adelaide
  - Monash Children's Hospital, Clayton, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia
- Canada (14):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - Children's & Women's Health Centre of British Columbia, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Izaak Walton Killam (IWK) Health Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital, London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - CHU de Québec - Université Laval, Québec, Quebec
  - CHU de Sherbrooke, Sherbrooke, Quebec
  - Saskatchewan Health Authority, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No